CLINICAL TRIAL: NCT05225155
Title: Effect of Prophylatic Use of Enoxaparin in Women Undergoing in Vitro Fertilization Treatment
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Luciano de Melo Pompei', Auxiliary Professor at Gynecology Department, Faculdade de Medicina do ABC
Other Study IDs: 41006620.0.0000.0082
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female; Thrombophilia; Fertilization in Vitro
Keywords: female infertility; thrombophilia; enoxaparin; abortion; in vitro fertilization; low molecular weight heparin
MeSH Terms: conditions — Infertility, Female; Thrombophilia | interventions — Enoxaparin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control: Women without thrombophilia, submitted to in vitro fertilization techniques
- Untreated Thrombophilia: Women with laboratorial thrombophilia, submitted to in vitro fertilization techniques, without treatment with enoxaparin
- Treated Thrombophilia: Women with laboratorial thrombophilia, submitted to in vitro fertilization techniques, and treated with enoxaparin
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Women with thrombophilia were treated with 40 mg daily of enoxaparin (treated group), initiated on the day of embryo transfer, up to week 36 of gestation
  Groups: Treated Thrombophilia

SUMMARY:
Retrospective study designed to evaluate outcomes in patients undergoing assisted reproduction. Some of them had thrombophilia, and part of them was treated with enoxaparin, started on the day of embryo transfer, and the other part not. Women without thrombophilia formed the control group.

DETAILED DESCRIPTION:
A retrospective study was performed to evaluate the results in 104 patients undergoing to assisted reproduction. Women without thrombophilia were included as controls (n=20), while women with thrombophilia were either treated with 40 mg daily of enoxaparin (treated group, n=54), initiated on the day of embryo transfer, and continued to the week 36 of gestation, or did not receive this medication (untreated group, n= 30).

ELIGIBILITY:
Inclusion Criteria:

* Women with female infertility or unexplained infertility
* Normal sperm analysis

Exclusion Criteria:

* Women who did not agree with in vitro fertilization techniques

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All included patients underwent in vitro fertilization (IVF) treatment with intracytoplasmic sperm injection (ICSI). Patients were initially submitted to controlled ovarian hyperstimulation under a short protocol with gonadotropins and GnRH antagonist. Women with laboratorial thrombophilia could be treated or not with enoxaparin according to her physician's decision. Women without detectable thrombophilia formed the control group.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with detectable fetal heartbeat | Day 28
  A transvaginal ultrasound was performed for detection of fetal heartbeat
Number of participants with detectable ongoing pregnancy | Week 12
  Ongoing pregnancy was detected by ultrasound at twelve weeks
Number of participants who delivered a live baby | Week 36
  Live birth was considered delivery that resulted in at least one live born neonate

SECONDARY OUTCOMES:
Number of participants with biochemical gestation detected | Day 14
  Serum beta-HCG detected 14 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pompei, Study Director — Faculdade de Medicina do ABC
Locations (1):
- Assistencia Materno Infantil Lambert, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing was not approved yet by our ethical committee board